CLINICAL TRIAL: NCT00851565
Title: Use of Combined Measurements of Serum Infliximab and Anti-infliximab Antibodies in the Treatment of Patients With Crohns Disease Failing Infliximab Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Aase and Ejnar Danielsens Foundation (Other); Beckett Foundation (Other); the Danish Biotechnology Program (Unknown); Colitis-Crohn Foreningen (Other); Danish Medical Association (Other); Frode V. Nyegaard and wife's Foundation (Unknown); Health Science Research Foundation of Region of Copenhagen (Unknown); Herlev Hospital Research Council (Unknown); Lundbeck Foundation (Other); P. Carl Petersens Fund (Other); Biomonitor A/S (Unknown); Prometheus Inc. (Industry); The Danish Institute for Health Services Research (Unknown)
Responsible Party: Mark A. Ainsworth, M.D., Ph.D. DMSci, Department of Medical Gastroenterology, Copenhagen University Hospital Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01MA
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients with Crohn's disease with secondary loss of response to infliximab.
  Interventions: Procedure: Measurement of serum infliximab and anti-infliximab antibodies
- 2 (Active Comparator): Patients with Crohn's disease with secondary loss of response to infliximab.
  Interventions: Procedure: Treatment according to current standards without knowledge of serum infliximab and anti-infliximab Ab status

INTERVENTIONS:
Procedure: Measurement of serum infliximab and anti-infliximab antibodies — In the intervention group treatment of patients with Crohn's disease with secondary loss of response to infliximab is based on serum infliximab and anti-infliximab Ab levels according to following algorithm:
  1. Low s-infliximab in the presence of anti-infliximab Ab: Adalimumab 80 mg s.c. followed by 40 mg every 2 weeks.
  2. Low s-infliximab without anti-infliximab Ab: Infliximab 10 mg/kg i.v. every 8 weeks.
  3. High s-infliximab without anti-infliximab Ab: Stop infliximab treatment. Review history. Steroids or surgery.
  4. High s-infliximab in the presence of anti-infliximab Ab: Same as number 3.
  Arms: 1
Procedure: Treatment according to current standards without knowledge of serum infliximab and anti-infliximab Ab status — In the control group patients with Crohn's disease with secondary loss of response to infliximab is treated according to current standard of care which is to increase dose of infliximab to 5 mg/kg every 4 weeks without knowledge of serum infliximab levels and anti-infliximab Ab status.
  Arms: 2

SUMMARY:
To compare treatment outcome in patients with Crohn's disease with secondary loss of response to infliximab (i.e. initial good response follow by loss of response) treated according to current standards based only on clinical features versus treatment based on serum levels of infliximab and anti-infliximab antibody (Ab) status.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand the information given to him/her and give written informed consent.
2. Definitive diagnosis of Crohn's disease (confirmed by recent radiological, endoscopic and/or histological evidence according to international criteria) .
3. Age minimum 18 years.
4. Previous good response to at least 3 doses (5mg/kg) of infliximab (as judged by the treating physician).
5. Loss of response to standard doses of infliximab (as judged by the treating physician).
6. Last infliximab infusion given at least 4 weeks before inclusion.
7. For patients with luminal disease, the CDAI should be above 220 points at inclusion.
8. For patients with fistulising disease only, at least one draining perianal fistula (confirmed by radiography, MR, ultrasound or physical examination) should be present.

Exclusion Criteria:

1. Any contraindication to continued infliximab treatment
2. Short bowel syndrome
3. Bowel resection within 12 weeks of inclusion.
4. Current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
5. Pregnancy
6. History of alcohol or drug abuse within the prior year
7. Patients who do not meet concomitant medication criteria.
8. Any other condition, which in the Investigator's judgment would make the patient unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with response at week 12, i.e. CDAI decrease of 70 or more for patients with luminal disease, or reduction of 50 percent or more from base line in the number of draining fistulas for patients with fistulising disease. | 12 weeks
  Clinical response rates at week 12 should be non-inferior in the intervention group as compared to the control group.
  Both primary end-points should be met in order to declare the primary end-points succesfully archived.
Total expenses related to Crohn's disease during the study (inclusion to week 12). | 12 weeks
  Crohn related expenses at week 12 should be less in the intervention group as compared to the control group.
  Both primary end-points should be met in order to declare the primary end-points succesfully archived.

SECONDARY OUTCOMES:
Mean change compared to baseline in WPAI score at week 12. | 12 weeks
Mean change compared to baseline in IBDQ score at week 12. | 12 weeks
Mean change compared to baseline in CDAI score at week 4,8, 12,20. | 4, 8, 12, 20 weeks
Mean change compared to baseline in PDAI score at week 4, 8, 12, and 20. | 4, 8, 12, 20 weeks
Clinical response at week 4, 8, 20 | Week 4, 8, 20
  Clinical response is defined as decrease of 70 in CDAI (luminal disease) or 50% reduction of active fistulas (fistulizing disease).
Laboratory parameters | Week 12
  Change in laboratory parameters (hemoglobin, crp, albumin) from inclusion to week 12.
Days with subjective feeling of disability due to Crohn's disease | week 12
  Total number of days with subjective feelinhg of disability due to Crohn's disease from inclusion to week 12.
Serious adverse drug reactions | week 12
  Total number of serious adverse drug reactions from inclusion to week 12.
Expenses related to Crohn's diseae at week 20 | week 20
Expenses related to Crohn's disease compared to change in CDAI-score (luminal disease) or PDAI-score (fistulizing disease), and IBD-score at week 12 and 20 | week 12 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ainsworth, M.D., Ph.D. DMSci, Principal Investigator
Locations (8):
- Denmark (8):
  - Dept of Medical Gastroenterology, Ålborg University Hospital, Aalborg
  - Dept of Hepatology and Medical Gastroenterology, Århus University Hospital, Aarhus
  - Institute for Inflammation Research, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Herlev University Hospital, Herlev
  - Department of Gastroenterology, Hvidovre University Hospital, Hvidovre
  - Department of Medical Gastroenterology, Køge University Hospital, Køge
  - Dept of Medical Gastroenterology, Odense University Hospital, Odense

REFERENCES:
- [Background] Ainsworth MA, Bendtzen K, Brynskov J. Tumor necrosis factor-alpha binding capacity and anti-infliximab antibodies measured by fluid-phase radioimmunoassays as predictors of clinical efficacy of infliximab in Crohn's disease. Am J Gastroenterol. 2008 Apr;103(4):944-8. doi: 10.1111/j.1572-0241.2007.01638.x. Epub 2007 Nov 19. PMID 18028512
- [Background] Bendtzen K, Ainsworth M, Steenholdt C, Thomsen OO, Brynskov J. Individual medicine in inflammatory bowel disease: monitoring bioavailability, pharmacokinetics and immunogenicity of anti-tumour necrosis factor-alpha antibodies. Scand J Gastroenterol. 2009;44(7):774-81. doi: 10.1080/00365520802699278. PMID 19140087
- [Background] Bendtzen K, Geborek P, Svenson M, Larsson L, Kapetanovic MC, Saxne T. Individualized monitoring of drug bioavailability and immunogenicity in rheumatoid arthritis patients treated with the tumor necrosis factor alpha inhibitor infliximab. Arthritis Rheum. 2006 Dec;54(12):3782-9. doi: 10.1002/art.22214. PMID 17133559
- [Background] Svenson M, Geborek P, Saxne T, Bendtzen K. Monitoring patients treated with anti-TNF-alpha biopharmaceuticals: assessing serum infliximab and anti-infliximab antibodies. Rheumatology (Oxford). 2007 Dec;46(12):1828-34. doi: 10.1093/rheumatology/kem261. PMID 18032541
- [Derived] Steenholdt C, Brynskov J, Thomsen OO, Munck LK, Christensen LA, Pedersen G, Kjeldsen J, Ainsworth MA. Implications of Infliximab Treatment Failure and Influence of Personalized Treatment on Patient-reported Health-related Quality of Life and Productivity Outcomes in Crohn's Disease. J Crohns Colitis. 2015 Nov;9(11):1032-42. doi: 10.1093/ecco-jcc/jjv139. Epub 2015 Aug 5. PMID 26245216
- [Derived] Steenholdt C, Bendtzen K, Brynskov J, Thomsen OO, Munck LK, Christensen LA, Pedersen G, Kjeldsen J, Ainsworth MA. Changes in serum trough levels of infliximab during treatment intensification but not in anti-infliximab antibody detection are associated with clinical outcomes after therapeutic failure in Crohn's disease. J Crohns Colitis. 2015 Mar;9(3):238-45. doi: 10.1093/ecco-jcc/jjv004. Epub 2015 Jan 9. PMID 25576753
- [Derived] Steenholdt C, Brynskov J, Thomsen OO, Munck LK, Fallingborg J, Christensen LA, Pedersen G, Kjeldsen J, Jacobsen BA, Oxholm AS, Kjellberg J, Bendtzen K, Ainsworth MA. Individualised therapy is more cost-effective than dose intensification in patients with Crohn's disease who lose response to anti-TNF treatment: a randomised, controlled trial. Gut. 2014 Jun;63(6):919-27. doi: 10.1136/gutjnl-2013-305279. Epub 2013 Jul 22. PMID 23878167